CLINICAL TRIAL: NCT00328536
Title: Effects of Treatment With Omacor for 6 Weeks on Preprandial and Postprandial Endothelial Function Following a High Fat Meal in Patients With Type 2 Diabetes Mellitus
Brief Title: Omacor for the Treatment of Vascular Dysfunction in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Heart and Diabetes Center North-Rhine Westfalia (Other); Solvay Pharmaceuticals (Industry)
Responsible Party: Heart and Diabetes Center, Diabetes Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OMACOR-D-01/06
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Atherosclerosis; Type 2 Diabetes Mellitus
Keywords: flow-mediated vasodilatation; endothelial dysfunction; omega-3 fatty acids; type 2 diabetes mellitus; postprandial state
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2 | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Omacor

SUMMARY:
The purpose of the study is to determine whether a 6-week treatment with 4 g Omacor/day improves the baseline and postprandial endothelial function (after a high-fat meal) in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus (T2DM) have a 2 to 5-fold increase in cardiovascular mortality compared to non-diabetics.

Endothelial dysfunction (ED) is an early messenger of atherosclerosis and is present in states showing a high cardiovascular (CV) risk, such as active and passive smoking, dyslipidemia, arterial hypertension, obesity, hyperhomocysteinemia, coronary artery disease, congestive heart failure and type 1 and type 2 diabetes mellitus. Endothelial function is a variable with a large day-to-day variation and shows great excursions even within one day. Several factors might play a role such as hormonal status, physical activity, sleep quality, but the most important seems to be the postprandial state. Postprandial ED was demonstrated not only in patients with CV disease or diabetes, but even in healthy subjects. A large body of evidence has accumulated showing distinctive and cumulative effects of hyperglycemia and hypertriglyceridemia on postprandial ED. Since postprandial dysmetabolism was linked to CVD, ED was proposed to be the mechanism connecting them. Considering that the postprandial state covers most of our daytime, interventions targeting a reduction in postprandial ED might play a decisive role in atherosclerosis prevention.

For the treatment of postprandial ED several therapeutical approaches have been suggested such as folic acid, tetrahydrobiopterin, vitamins C and E and statins.

Some properties of omega-3 fatty acids suggest that such an impairment of postprandial endothelial dysfunction could be prevented by treatment with Omacor® and the purpose of our study is to demonstrate that a six-week therapy with Omacor prevents endothelial dysfunction in fasting state and following a high-fat meal.

Several controlled clinical studies conducted in persons with TM2DM or after myocardial infarction have shown that consumption of omega-3 long chain polyunsaturated fatty acids (n-3 PUFA) have several beneficial effects such as: lowers risk of primary cardiac arrest, reduces triglyceride levels, increases high-density lipoprotein levels, reduces platelet aggregability, acts anti-inflammatory and immune-modulating, lowers blood pressure and improves endothelial function.

Consumption of n-3 fatty acids was shown to positively influence platelet, fibrinolytic and vascular function in hypertensive type 2 diabetic patients. Mediterranean- style diet restores markers of endothelial dysfunction and inflammation in persons with metabolic syndrome and improves endothelial function in hypercholesterolemic men.

Since Omacor contains in high-dose purified n-3 fatty acids eicosapentaenoic and docosahexaenoic acid (EPA and DHA), our first hypothesis is that a 6-week therapy with 4g/d Omacor improves fasting endothelial function in persons with T2DM.

In patients with T2DM, a three-week diet with a high amount of polyunsaturated fatty acids compared to a diet with a high amount of monounsaturated fatty acids, produces a significantly lower increase in postprandial lipemia after an oral fat load. Since postprandial lipemia induces transient endothelial dysfunction, our second hypothesis is that treatment with Omacor prevents postprandial impairment of endothelial function after a high fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus

Exclusion Criteria:

* History of myocardial infarction, stroke
* Severe diabetes complications
* Severe hypo- or hypertension
* Chronic alcohol abuse
* Renal failure

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Postprandial (2, 4 and 6 hours) flow-mediated vasodilation after a 6-week treatment with Omacor

SECONDARY OUTCOMES:
Baseline flow-mediated vasodilation after a 6-week treatment with Omacor

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Tschoepe, MD, Prof., Principal Investigator — Heart and Diabetes Center North-Rhine Westfalia; Alin Stirban, MD, Principal Investigator — Heart and Diabetes Center North-Rhine Westfalia
Locations (1):
- Heart- and Diabetes Centre NRW, Diabetes Clinic, Bad Oeynhausen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Stirban A, Nandrean S, Gotting C, Stratmann B, Tschoepe D. Effects of n-3 polyunsaturated fatty acids (PUFAs) on circulating adiponectin and leptin in subjects with type 2 diabetes mellitus. Horm Metab Res. 2014 Jun;46(7):490-2. doi: 10.1055/s-0033-1363225. Epub 2013 Dec 19. PMID 24356795